CLINICAL TRIAL: NCT01804270
Title: A Randomized, Double-Blinded, Sham-Controlled Trial of Repetitive Transcranial Magnetic Stimulation in Depressed Adolescents
Brief Title: rTMS for Depressed Teens: A Sham-Controlled Trial, Part 1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study & IDE was converted to Industry held, as opposed to initial investigator held.
Sponsor: Paul E. Croarkin (Other)
Responsible Party: Sponsor-Investigator, Paul E. Croarkin, Assistant Professor of Child and Adolescent Psychiatry, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-003248 Part 1
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Major Depressive Disorder
Keywords: Teen; Adolescent; Depression; Transcranial Magnetic Stimulation; TMS
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Part 1 Active (Active Comparator): Blinded, active repetitive transcranial magnetic stimulation
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- Part 1 Sham (Sham Comparator): Blinded, sham repetitive transcranial magnetic stimulation
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — Active treatments with repetitive transcranial magnetic stimulation (rTMS) consists of treatment settings of 120% magnetic field intensity relative to the patient's resting motor threshold, at 10 pulses per second (10 Hz) for 4 seconds, with an intertrain interval of 26 seconds for a total of 75 trains per treatment session.
  Other Names: NeuroStar XPLOR

SUMMARY:
This research proposal aims to better understand the neurobiology of depression in adolescents and how repetitive transcranial magnetic stimulation (rTMS) may therapeutically impact brain function and mood. This study will be the first to use a randomized, double-blinded, sham-controlled approach to the investigation of rTMS therapy for depressed adolescents. This approach will allow for the validation of rTMS treatment outcomes in the depressed adolescent population in a scientifically rigorous manner. The magnetic resonance (MR) spectroscopy pattern of rTMS response will be analyzed according to previously established protocols.

DETAILED DESCRIPTION:
Part 1 of the study aims to:

* Evaluate the antidepressant effects of daily, active rTMS (when compared with sham treatment) in adolescents meeting criteria for Major Depressive Disorder, single or recurrent episode.
* Evaluate, by proton magnetic resonance spectroscopy (1H-MRS) at 3 Tesla(3T), neurometabolic biomarkers at the beginning and end of each study phase.

  * Define regional specificity [anterior cingulate (AC) and left dorsolateral prefrontal cortex (L-DLPFC)] of cerebral metabolites(i.e. glutamate and glutamine) in adolescent depression.
  * Study whether specific neurochemical resonances are associated with response, remission, and/or maintenance of improvement of clinical depressive symptoms when rTMS is used to treat adolescent depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unipolar major depressive disorder, in a current major depressive episode, without psychotic features
* Pretreatment CDRS-R Raw score ≥ 40
* Age is at least 12 and less than 22 years
* Ongoing, stable dose antidepressant therapy for at least 6 weeks to include the following antidepressants (with dosing range):

  * Celexa (citalopram hydrobromide) - 10 to 60mg
  * Cymbalta (duloxetine) - 40mg to 120mg
  * Desyrel (trazodone HCl) - 12.5mg to 150mg
  * Effexor (venlafaxine HCl) - 37.5mg to 300mg
  * Luvox (fluvoxamine maleate) - 25mg to 200mg
  * Lexapro (escitalopram oxalate) - 10mg to 40mg
  * Paxil (paroxetine HCl) - 10mg to 50mg
  * Pristiq (desvenlafaxine) - 50mg to 100mg
  * Prozac (fluoxetine HCl) - 10mg to 80mg
  * Remeron (mirtazapine) - 7.5mg to 45mg
  * Savella (milnacipran HCl) - 25mg to 200mg
  * Zoloft (sertraline HCl) - 25mg to 200mg
* Subjects able to attend at least 31 study visits at study site.
* Willing to provide informed assent (adolescent) and informed consent (family)

Exclusion Criteria:

* Subjects currently on stimulant, antipsychotic, bupropion or tricyclic antidepressant medications.
* Prior rTMS, vagus nerve stimulation (VNS) or electroconvulsive therapy (ECT)
* Contraindication to MRI
* Contraindication to rTMS (history of neurological disorder such as seizures, increased intracranial pressure, brain surgery, or head trauma with loss of consciousness for >15 minutes, history of stroke, family history of epilepsy, intracardiac lines, Anticoagulant, immune suppressive and/or chemotherapy, or those who received any of these therapies within 3 months before enrollment in the study Unstable medication conditions such as hematological or infectious (e.g., human immunodeficiency virus-HIV) disorders, implanted electronic device, metal in the head, or pregnancy)
* History of schizophrenia, schizoaffective disorder, other [non mood disorder] psychosis, depression secondary to a medical condition, mental retardation, substance dependence or abuse within the past year (except nicotine), bipolar disorder, psychotic features in this or previous episodes, amnestic disorder, obsessive compulsive disorder, post-traumatic stress disorder, panic disorder
* History of autoimmune, endocrine, viral, or vascular disorder.
* Unstable cardiac disease, uncontrolled hypertension, or sleep apnea
* Active suicidal intent or plan, or history of attempt within the past 6 months

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Croarkin, DO, Principal Investigator — Mayo Clinic; Mark A George, MD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Sonmez AI, Kucuker MU, Lewis CP, Kolla BP, Doruk Camsari D, Vande Voort JL, Schak KM, Kung S, Croarkin PE. Improvement in hypersomnia with high frequency repetitive transcranial magnetic stimulation in depressed adolescents: Preliminary evidence from an open-label study. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Mar 8;97:109763. doi: 10.1016/j.pnpbp.2019.109763. Epub 2019 Oct 18. PMID 31634515
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1 Active | Part 1 Sham
Started | 2 | 4
Completed | 1 | 3
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Active | Part 1 Sham | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (1.41) | 17.25 (1.5) | 16.5 (1.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Children's Depression Rating Scale-Revised (CDRS-R) Post Treatment 30 or Last Treatment (in the Case of Early Withdrawal)
Description: The Children's Depression Rating Scale-Revised (CDRS-R) is a validated, 17-item, semi-structured clinician rating tool to assess severity of depression with subject and parental input for 14 of the 17 items.
Time Frame: Within 5 days after Treatment 30 or Last Treatment
Population: Terminated study. Data was not collected nor analyzed
Arm/Group | Part 1 Active | Part 1 Sham
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Mean Change From Baseline in Clinical Global Impression - Severity (CGI-S) Post Treatment 30 or Last Treatment (in the Case of Early Withdrawal)
Description: The Clinical Global Impression - Severity (CGI-S) is a standardized assessment utilizing a 7-point scale with which the clinician rates the severity of the subject's depressive illness at the time of assessment relative to the clinician's past experience with patients who have the same diagnosis.
Time Frame: Within 5 days after Treatment 30 or Last Treatment
Population: Terminated study. Data was not collected nor analyzed.
Arm/Group | Part 1 Active | Part 1 Sham
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Mean Clinical Global Impression - Improvement (CGI-I) Score Post Treatment 30 or Last Treatment (in the Case of Early Withdrawal)
Description: The Clinical Global Impression - Improvement (CGI-I) is a standardized assessment utilizing a 7-point scale with which the clinician rates the degree to which the severity of the subject's depressive illness has improved or worsened compared to baseline severity.
Time Frame: Within 5 days after Treatment 30 or Last Treatment
Population: Terminated study. Data was not collected nor analyzed.
Arm/Group | Part 1 Active | Part 1 Sham
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 6 months.
Arm/Group | Part 1 Active | Part 1 Sham
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/4
Other Adverse Events (participants affected / at risk) | 2/2 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Active (N=2) | Part 1 Sham (N=4)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Active (N=2) | Part 1 Sham (N=4)
Headaches (Nervous system disorders) | 2 (15) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT01804270/Prot_SAP_000.pdf